CLINICAL TRIAL: NCT01973036
Title: Foley Catheter Versus Oxytocin for Labor Induction in Women With Term and Near Term Premature Rupture of Membranes: A Randomized Clinical Trial (FOLCROM Trial)
Brief Title: FOLCROM Trial: Foley Catheter in Rupture of Membranes
Acronym: FOLCROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0379
Record Dates: First submitted 2013-09-17; First posted 2013-10-31 (Estimated); Results first posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-07

CONDITIONS: Premature Rupture of Membranes
Keywords: foley catheter; foley bulb; oxytocin
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Active Comparator): This arm will receive oxytocin at a rate of 2 milliunits/milliliter. If the fetal status is reassuring, this can be increased by 2 milliunits/milliliter every 30 minutes to achieve an adequate contraction pattern as per the institution's definition to a maximum of 30 milliunits/milliliter. This infusion may be continued until delivery.
  Interventions: Drug: Oxytocin
- Foley Catheter and Oxytocin (Experimental): A 30cc/16 French (16F) foley catheter will be inserted by the provider under direct visualization or by palpation, ensuring that the catheter is appropriately and adequately positioned. Oxytocin will be administered concurrently at a rate of 2 milliunits/milliliter (as noted under oxytocin active comparator). If the catheter remains in place after 12 hours, it will be deflated and removed and oxytocin infusion will continue.
  Interventions: Device: Foley Catheter; Drug: Oxytocin

INTERVENTIONS:
Device: Foley Catheter — The balloon will be inflated with 30 cc of sterile saline. The catheter will be taped to the patient's leg so that traction is maintained. The catheter will be assessed hourly for expulsion by a health care provider by applying gentle traction on the catheter or a vaginal examination if it is unclear by traction. Once the Foley catheter is expelled or 12 hours reached, the induction will be continued with oxytocin per this protocol.
  Other Names: 30cc/16 French
  Arms: Foley Catheter and Oxytocin
Drug: Oxytocin — Each arm will receive oxytocin at a rate of 2 milliunits/milliliter. If the fetal status is reassuring, this can be increased by 2 milliunits/milliliter every 30 minutes to achieve an adequate contraction pattern as per the institution's definition to a maximum of 30 milliunits/milliliter. This infusion may be continued until delivery.
  Other Names: Pitocin

SUMMARY:
Multicenter randomized clinical trial comparing oxytocin versus oxytocin and foley catheter for induction in women who present with premature rupture of membranes who are not in labor.

DETAILED DESCRIPTION:
This is a prospective, randomized, multi-center clinical trial to test the hypothesis that in women with term and near term premature rupture of membranes (PROM), an intrauterine Foley catheter plus oxytocin infusion will decrease the mean time from induction to delivery by 2.5 hours as compared to oxytocin alone.

ELIGIBILITY:
Inclusion Criteria:

1. Spontaneous rupture of membranes (ROM) ≥1 hour prior to starting induction; ROM defined as clinical history with the presence of 2 of the following 4: pooling, ferning, nitrazine, oligohydramnios. In the absence of clinical history, oligohydramnios AND pooling must be present for ROM to be diagnosed. Oligohydramnios is defined as a total amniotic fluid index of <5cm or a maximum vertical pocket <2cm.
2. Unfavorable cervix, defined as sterile digital exam ≤ 2cm dilated / 80% effaced
3. Gestational age ≥ 34 weeks by best obstetric estimate
4. Clinical management decision is vaginal delivery
5. Singleton gestation
6. Cephalic presentation
7. Willing to participate and able to understand and sign the informed consent document before randomization
8. Women of reproductive age

Exclusion Criteria:

1. Multiple gestations
2. Lethal fetal anomalies, e.g., anencephaly, trisomy 13, trisomy 18
3. Latex allergy
4. Greater than 1 prior cesarean delivery
5. Active labor - defined as contractions more frequent than every 5 minutes (or ≥ 12 contractions in 1 hour) associated with ≥ 1 cm cervical change. In the absence of ≥ 1 cm cervical change after 2 hours, patients with contractions can be included in the study.
6. Suspicion of chorioamnionitis
7. Any contraindications to vaginal delivery, including malpresentation, active herpes, complete placenta previa, greater than two prior cesarean deliveries, etc.
8. HIV positive status or AIDS
9. Intrauterine fetal demise
10. Suspected placental abruption, significant hemorrhage
11. Nonreassuring fetal heart rate (FHR) pattern
12. Participation in a competing trial

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Awathif D Mackeen, MD, MPH, Principal Investigator — Geisinger Clinic
Locations (5):
- United States (5):
  - Banner Good Samaritan Regional Medical Center, Phoenix, Arizona
  - Christiana Care Health System CCHS, Newark, Delaware
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ACOG Practice Bulletin No. 107: Induction of labor. Obstet Gynecol. 2009 Aug;114(2 Pt 1):386-397. doi: 10.1097/AOG.0b013e3181b48ef5. No abstract available. PMID 19623003
- [Background] Gunn GC, Mishell DR Jr, Morton DG. Premature rupture of the fetal membranes. A review. Am J Obstet Gynecol. 1970 Feb 1;106(3):469-83. doi: 10.1016/0002-9378(70)90378-9. No abstract available. PMID 4905833
- [Background] LANIER LR Jr, SCARBROUGH RW Jr, FILLINGIM DW, BAKER RE Jr. INCIDENCE OF MATERNAL AND FETAL COMPLICATIONS ASSOCIATED WITH RUPTURE OF THE MEMBRANES BEFORE ONSET OF LABOR. Am J Obstet Gynecol. 1965 Oct 1;93:398-404. doi: 10.1016/0002-9378(65)90068-2. No abstract available. PMID 14337377
- [Background] Lin MG, Nuthalapaty FS, Carver AR, Case AS, Ramsey PS. Misoprostol for labor induction in women with term premature rupture of membranes: a meta-analysis. Obstet Gynecol. 2005 Sep;106(3):593-601. doi: 10.1097/01.AOG.0000172425.56840.57. PMID 16135593
- [Background] Wolff K, Swahn ML, Westgren M. Balloon catheter for induction of labor in nulliparous women with prelabor rupture of the membranes at term. A preliminary report. Gynecol Obstet Invest. 1998;46(1):1-4. doi: 10.1159/000009986. PMID 9692332
- [Result] Boulvain M, Kelly A, Lohse C, Stan C, Irion O. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2001;(4):CD001233. doi: 10.1002/14651858.CD001233. PMID 11687101
- [Result] Hannah ME, Ohlsson A, Farine D, Hewson SA, Hodnett ED, Myhr TL, Wang EE, Weston JA, Willan AR. Induction of labor compared with expectant management for prelabor rupture of the membranes at term. TERMPROM Study Group. N Engl J Med. 1996 Apr 18;334(16):1005-10. doi: 10.1056/NEJM199604183341601. PMID 8598837
- [Result] Fitzpatrick CB, Grotegut CA, Bishop TS, Canzoneri BJ, Heine RP, Swamy GK. Cervical ripening with foley balloon plus fixed versus incremental low-dose oxytocin: a randomized controlled trial. J Matern Fetal Neonatal Med. 2012 Jul;25(7):1006-10. doi: 10.3109/14767058.2011.607522. Epub 2011 Dec 14. PMID 21793769
- [Result] Pettker CM, Pocock SB, Smok DP, Lee SM, Devine PC. Transcervical Foley catheter with and without oxytocin for cervical ripening: a randomized controlled trial. Obstet Gynecol. 2008 Jun;111(6):1320-6. doi: 10.1097/AOG.0b013e31817615a0. PMID 18515515
- [Result] Oliveira MV, Oberst PV, Leite GK, Aguemi A, Kenj G, Leme VD, Sass N. [Cervical Foley catheter versus vaginal misoprostol for cervical ripening and induction of labor: a randomized clinical trial]. Rev Bras Ginecol Obstet. 2010 Jul;32(7):346-51. doi: 10.1590/s0100-72032010000700007. Portuguese. PMID 21152844
- [Result] Sanchez-Ramos L, Chen AH, Kaunitz AM, Gaudier FL, Delke I. Labor induction with intravaginal misoprostol in term premature rupture of membranes: a randomized study. Obstet Gynecol. 1997 Jun;89(6):909-12. doi: 10.1016/s0029-7844(97)00113-0. PMID 9170463
- [Result] Wing DA, Paul RH. Induction of labor with misoprostol for premature rupture of membranes beyond thirty-six weeks' gestation. Am J Obstet Gynecol. 1998 Jul;179(1):94-9. doi: 10.1016/s0002-9378(98)70256-x. PMID 9704771
- [Result] Zeteroglu S, Engin-Ustun Y, Ustun Y, Guvercinci M, Sahin G, Kamaci M. A prospective randomized study comparing misoprostol and oxytocin for premature rupture of membranes at term. J Matern Fetal Neonatal Med. 2006 May;19(5):283-7. doi: 10.1080/14767050600589807. PMID 16753768
- [Result] Tan PC, Daud SA, Omar SZ. Concurrent dinoprostone and oxytocin for labor induction in term premature rupture of membranes: a randomized controlled trial. Obstet Gynecol. 2009 May;113(5):1059-1065. doi: 10.1097/AOG.0b013e3181a1f605. PMID 19384121
- [Derived] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2023 Mar 30;3(3):CD001233. doi: 10.1002/14651858.CD001233.pub4. PMID 36996264
- [Derived] Mackeen AD, Durie DE, Lin M, Huls CK, Qureshey E, Paglia MJ, Sun H, Sciscione A. Foley Plus Oxytocin Compared With Oxytocin for Induction After Membrane Rupture: A Randomized Controlled Trial. Obstet Gynecol. 2018 Jan;131(1):4-11. doi: 10.1097/AOG.0000000000002374. PMID 29215519

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women presenting to labor & delivery with ruptured membranes with an unfavorable cervix based on sterile digital exam at greater than or equal to 34 weeks were approached by a study team member for participation.
Groups:
- Foley Catheter and Oxytocin: Foley Catheter: A 30cc/16 French (16F) foley catheter will be inserted. Balloon will be inflated with 30 cc of sterile saline. The catheter will be taped to the patient's leg so that traction is maintained. The catheter will be assessed hourly for expulsion by a health care provider by applying gentle traction on the catheter or a vaginal examination if it is unclear by traction. Once the Foley catheter is expelled or 12 hours reached, the induction will be continued with oxytocin per this protocol.
  Oxytocin: administered concurrently at a rate of 2 milliunits/milliliter. If the fetal status is reassuring, this can be increased by 2 milliunits/milliliter every 30 minutes to achieve an adequate contraction pattern as per the institution's definition to a maximum of 30 milliunits/milliliter. This infusion may be continued until delivery.
Period: Overall Study
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Started (The group to which the subject was randomized) | 108 | 93
Received Assigned Intervention (The intervention completed. (Some subjects rejected arm assignment or required opposite treatment.)) | 113 | 88
Completed (Data analyzed according to original arm assignment, not treatment completed.) | 108 | 93
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Foley Catheter and Oxytocin: A 30cc/16 French (16F) foley catheter will be inserted by the provider under direct visualization or by palpation, ensuring that the catheter is appropriately and adequately positioned. Oxytocin will be administered concurrently at a rate of 2 milliunits/milliliter (as noted under oxytocin active comparator). If the catheter remains in place after 12 hours, it will be deflated and removed and oxytocin infusion will continue.
  Foley Catheter: Balloon will be inflated with 30 cc of sterile saline. The catheter will be taped to the patient's leg so that traction is maintained. The catheter will be assessed hourly for expulsion by a health care provider by applying gentle traction on the catheter or a vaginal examination if it is unclear by traction. Once the Foley catheter is expelled or 12 hours reached, the induction will be continued with oxytocin per this protocol.
  Oxytocin: Each arm will receive oxytocin at a rate of 2 milliunits/milliliter. If the fetal status is reassuri
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Foley Catheter and Oxytocin | Total
Number analyzed (Participants) | 108 | 93 | 201
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [22.8 to 31.4] | 27.5 [23.4 to 32.2] | 27.25 [23.35 to 31.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 93 | 201
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time From Induction of Labor Until Delivery
Description: Time from induction (i.e., start time of Foley catheter or oxytocin) to delivery (hours), analyzed for all deliveries
Time Frame: Time from induction to delivery (average 14.2 hours)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 108 | 93
hours | 14.4 (7.9) | 13.9 (6.9)

2. Secondary Outcome: Number of Participants With Chorioamnionitis
Description: Number of participants with chorioamnionitis excluding all those who were hospitalized with preterm premature rupture of membranes (PPROM) prior to 34 0/7 weeks. Chorioamnionitis was defined as temperature 38°C (or 100.4°F) or greater with at least two of the following: purulent discharge, maternal tachycardia (heart rate 100 beats per minute or greater), fetal tachycardia (heart rate 160 beats per minute or greater), foul odor of the amniotic fluid, or maternal leukocytosis (greater than 15,000 cells/mL3).
  Without Restriction = Chorioamnionitis was defined as temperature 38°C or greater and one of the following: purulent discharge, maternal tachycardia, fetal tachycardia, foul odor of the amniotic fluid, or maternal leukocytosis.
  With Restriction = Chorioamnionitis was defined as temperature 38°C or greater and two of the following: purulent discharge, maternal tachycardia, fetal tachycardia, foul odor of the amniotic fluid, or maternal leukocytosis.
Time Frame: Duration of Labor (average 4.8 hours)
Population: The number of participants analyzed excludes patients who were hospitalized with PPROM prior to 34 0/7 weeks (i.e., four patients in the Oxytocin arm and six patients in the Foley Catheter arm).
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 104 | 87
Participants
  Without Restrictions | 2 | 9
  With Restrictions | 0 | 7

3. Secondary Outcome: Number of Participants With Vaginal Delivery Within 12 Hours From Placement of Foley Catheter or Start Time of Oxytocin
Time Frame: Duration of Labor (average 4.8 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 108 | 93
Participants | 46 | 34

4. Secondary Outcome: Number of Participants With Vaginal Delivery Within 24 Hours From Placement of Foley Catheter or Start Time of Oxytocin
Time Frame: Duration of Labor (average 4.8 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 108 | 93
Participants | 80 | 61

5. Secondary Outcome: Duration of First, Second and Third Stage of Labor (Minutes) for Those Undergoing Vaginal Deliveries
Time Frame: Duration of Labor (average 4.8 hours)
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 80 | 61
Minutes
  First Stage | 130 [76.5 to 226] | 188 [111 to 294]
  Second Stage | 39 [15 to 88] | 23 [11 to 72]
  Third Stage | 5 [3 to 6] | 5 [3 to 7]

6. Secondary Outcome: Rate of Failed Induction of Labor as the Indication for Cesarean
Description: This will be defined by a combination of provider documentation and cervical dilation of ≤4cm/90% effaced or ≤5cm/any effacement after a minimum of 12 hours of oxytocin in the setting of adequate contraction.
  One patient was missing information for failed induction.
Time Frame: Duration of Labor (average 4.8 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 21 | 25
Participants | 6 | 8

7. Secondary Outcome: Rate of Endomyometritis
Description: Endomyometritis defined as: Temperature ≥100.4°F + one of the following: fundal tenderness, maternal tachycardia (Heart Rate ≥ 100 BPM), purulent cervical discharge and no other source of fever
Time Frame: Duration of hospital stay (average 3.4 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 108 | 93
Participants | 0 | 0

8. Secondary Outcome: Maternal Length of Stay, From Admission to Discharge (Days)
Time Frame: Duration of hospital stay (average 3.4 days)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 108 | 93
days | 3 [2 to 3] | 3 [2 to 4]

9. Secondary Outcome: Rate of Five Minute Apgar Score < 5
Description: Apgar is a test for assessing a newborn shortly after birth to determine if extra medical care or emergency care may be needed. Usually administered at 1 and 5 minutes after birth, the test includes assessment of Appearance, Pulse, Grimace, Activity and Respiration. Scores range from 0 - 10.
Time Frame: Duration of hospital stay (average 3.4 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 108 | 93
Participants | 1 | 1

10. Secondary Outcome: Arterial Cord Blood Gas (pH), When Obtained
Time Frame: Within 1 hour of delivery
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 108 | 93
pH | 7.25 (0.07) | 7.26 (0.07)

11. Secondary Outcome: Rate of Neonatal Sepsis
Description: Neonatal sepsis [positive blood or cerebrospinal fluid (CSF) cultures]
Time Frame: Duration of hospital stay (average 3.4 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 108 | 93
Participants | 0 | 0

12. Secondary Outcome: Neonatal Intensive Care Unit (NICU) Admission Rate
Time Frame: Duration of hospital stay (average 3.4 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 108 | 93
Participants | 20 | 21

13. Secondary Outcome: Neonatal Length of Stay
Time Frame: Duration of hospital stay (average 3.4 days)
Measure: Median (Standard Deviation); unit: hours
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 108 | 93
hours | 49.7 (16.9) | 52.4 (20.0)

14. Secondary Outcome: Number of Participants With Confirmed Histologic Chorioamnionitis/Funisitis
Description: Chorioamnionitis/funisitis as determined by the pathologist examining the placenta
Time Frame: Duration of hospital stay (average 3.4 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 108 | 93
Participants | 9 | 10

15. Secondary Outcome: Time From Induction to Delivery (Hours)
Description: Time from induction to delivery (hours) excluding all those who were hospitalized with PPROM prior to 34 0/7 weeks
Time Frame: Time from induction to delivery (average 14.2 hours)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 104 | 87
hours | 14.23 (8.19) | 14.16 (6.97)

16. Secondary Outcome: Overall Cesarean Delivery
Time Frame: Duration of hospital stay (average 3.4 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 108 | 93
Participants | 21 | 25

17. Secondary Outcome: Rate of Chorioamnionitis
Description: Chorioamnionitis defined as (Temperature greater than or equal to 100.4 degrees fahrenheit or 38 degrees celsius) with at least 2 of the following: uterine tenderness, maternal tachycardia (HR greater than or equal to 100 bpm), fetal tachycardia (HR greater than or equal to 160bpm), foul odor of the amniotic fluid, or maternal leukocytosis (greater than 15000 cells/cubic milliliter)
Time Frame: Duration of hospital stay (average 3.4 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 108 | 93
Participants | 0 | 7

18. Secondary Outcome: Maternal Length of Stay From Delivery to Discharge (Hours)
Time Frame: Duration of hospital stay (average 3.4 days)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
Number analyzed (Participants) | 108 | 93
hours | 48.1 [38.8 to 57.2] | 47.8 [41.2 to 58.7]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time of randomization to the time the baby is discharged.
Arm/Group | Oxytocin | Foley Catheter and Oxytocin
All-Cause Mortality (participants affected / at risk) | 0/108 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/93
Other Adverse Events (participants affected / at risk) | 0/108 | 0/93

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No